CLINICAL TRIAL: NCT06338241
Title: Clinical Study to Analyze the Osteogenic Action of a Osteogenic Action of a Biphasic Bioceramic With Statin in a Third Molar Extraction Model (Galibone+) in Bone Regeneration Following the Extraction of Impacted Mandibular Third Molars
Brief Title: Osteogenic Action of a Biphasic Bioceramic With Statin in a Third Molar Extraction Model
Acronym: Galibone
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mario Pérez Sayáns (Other)
Collaborators: Universidad de Murcia (Other)
Responsible Party: Sponsor-Investigator, Mario Pérez Sayáns, Principal investigator of ORALRES Group, University of Santiago de Compostela
Organization: University of Santiago de Compostela (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CPP2021-008391
Record Dates: First submitted 2024-03-20; First posted 2024-03-29 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Bone Loss; Regenerative Inflammation
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Durapatite; Simvastatin; Bio-Oss

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Galibone Group (Experimental): The Galibone+ experimental group includes participants receiving Galibone+ after impacted mandibular third molar extraction, testing its osteogenic properties. Galibone+ is prepared per manufacturer's instructions, potentially by immersing in sterile saline. Applied post-extraction into the socket using specialized instruments, it's compared to a control group receiving Bio-Oss, a standard xenograft material. Experimental group patients receive postoperative medications, including antibiotics and pain management. Follow-up assesses pain, inflammation, complications, and bone regeneration via radiological evaluation. Goal: Assess Galibone+'s efficacy in bone regeneration versus control.
  Interventions: Combination Product: Biphasic bioceramic of tricalcium phosphate and hydroxyapatite with simvastatin
- Control group (Active Comparator): The control group serves as an active comparator to the Galibone+ experimental group in this study. Participants undergo identical impacted mandibular third molar extraction procedures as the experimental group but receive a standard material, likely Bio-Oss, instead of Galibone+.
  Bio-Oss, a widely used xenograft material in dental surgeries, acts as a benchmark due to its osteoconductive properties. Applied post-extraction into the socket with specialized instruments, it provides a reference for comparing Galibone+'s efficacy. Patients in the control group receive postoperative medications as per the study protocol, including antibiotics and pain management. Follow-up assesses pain, inflammation, complications, and bone regeneration via radiological evaluation.
  Interventions: Other: Bovine Hydroxyapatite

INTERVENTIONS:
Combination Product: Biphasic bioceramic of tricalcium phosphate and hydroxyapatite with simvastatin — The intervention description for Galibone+ in the study involves the application of this substance to promote bone regeneration following the extraction of impacted mandibular third molars. Galibone is indicated to treat segmental and cavity bone loss, aesthetic repairs and bone augmentations (such as inlay or onlay grafts); to fill dental alveolar bone; for the placement of dental implants; for the stabilization of osteotomies and prostheses in dentistry.
  Other Names: Galibone
  Arms: Galibone Group
Other: Bovine Hydroxyapatite — The intervention description for Bio-Oss in the study involves the application of this standard material to promote bone regeneration following the extraction of impacted mandibular third molars. Bio-Oss is a commonly used xenograft material known for its osteoconductive properties.
  Other Names: Bio-Oss
  Arms: Control group

SUMMARY:
The clinical study aims to assess the osteogenic effects of Galibone+ in bone regeneration post-extraction of impacted mandibular third molars.

DETAILED DESCRIPTION:
With a focus on both clinical and radiological outcomes, the study seeks to compare the efficacy of Galibone+ against a standard material (Bio-Oss) through a double-blind, randomized split-mouth trial involving 30 patients. Variables including pain, inflammation, and post-surgical complications will be monitored during the initial seven-day follow-up, while bone volume reduction and mineral density will be evaluated radiographically over a six-month period. The study's findings promise to shed light on the potential of Galibone+ as a promising adjunct in enhancing bone regeneration following dental extractions, thereby advancing oral surgical practices and patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be of legal age.
* Participants must provide informed consent for participation in the study.
* Participants must require extraction of both impacted mandibular third molars.
* Both impacted molars must exhibit a similar level of complexity for extraction.
* Participants must have no history of infection in the impacted molars prior to extraction.
* Participants must not have any contraindications to undergoing oral surgical procedures (ASA I/II classification).

Exclusion Criteria:

* Participants with severe mental disorders that may impair their ability to provide informed consent or follow study instructions.
* Participants currently receiving medications contraindicated for dental extractions.
* Participants under the age of legal consent.
* Participants who have undergone head and neck radiotherapy within the past 18 months.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-02 (Actual); Primary Completion 2025-06-02 (Estimated); Study Completion 2025-09-02 (Estimated)

PRIMARY OUTCOMES:
Bone Regeneration_Reduction in radiolucent volume | A) Immediately after extraction B) 1 month. C) 3 months. D) 6 months
  This outcome measure involves assessing the degree of bone regeneration in the extraction socket following the extraction of impacted mandibular third molars. It will be evaluated through radiological imaging using CBCT scans at specified time points, including immediately post-extraction, at one month, three months, and six months post-extraction.
  Reduction in radiolucent volume within the extraction socket, indicating new bone formation (Hounsfield unit (HU)).
  High values mean more radiopacity and better regeneration.
Bone Regeneration_bone volume | A) Immediately after extraction B) 1 month. C) 3 months. D) 6 months
  This outcome measure involves assessing the degree of bone regeneration in the extraction socket following the extraction of impacted mandibular third molars. It will be evaluated through radiological imaging using CBCT scans at specified time points, including immediately post-extraction, at one month, three months, and six months post-extraction.
  Evaluation of bone volume within the extraction site over time (mm3). The increase in bone volume means better regeneration.
Bone Regeneration_bone density | A) Immediately after extraction B) 1 month. C) 3 months. D) 6 months
  This outcome measure involves assessing the degree of bone regeneration in the extraction socket following the extraction of impacted mandibular third molars. It will be evaluated through radiological imaging using CBCT scans at specified time points, including immediately post-extraction, at one month, three months, and six months post-extraction.
  Changes in bone density within the regenerated bone tissue (Hounsfield unit (HU)) High values mean more radiopacity and better regeneration.
Bone Regeneration_Fractal dimension | A) Immediately after extraction B) 1 month. C) 3 months. D) 6 months
  This outcome measure involves assessing the degree of bone regeneration in the extraction socket following the extraction of impacted mandibular third molars. It will be evaluated through radiological imaging using CBCT scans at specified time points, including immediately post-extraction, at one month, three months, and six months post-extraction.
  Evaluation of bone morphology within the extraction site over time analyzing the fractal dimension (FD) FD can vary between 1 and 2, with 1 being a very simple fractal dimension (such as a straight line) and 2 being a more complex fractal dimension (such as a completely irregular surface).

SECONDARY OUTCOMES:
Pain levels through visual analog scale | 24 hours, 48 hours, 72 hours, and 7 days
  Assessment of pain experienced by participants using a visual analog scale (VAS) at various time points post-extraction. It comprehends values between 0-10, where 10 is the worst situation.
Clinical Inflammation evaluating by presence/absence | 24 hours, 48 hours, 72 hours, and 7 days
  Evaluation of postoperative inflammation around the extraction site using clinical examination and assessment tools (presence/absence).
  The presence of inflammation means the worst prognosis.
Healing measured by healing index | 24 hours, 48 hours, 72 hours, and 7 days
  The healing progress will be assessed using the Healing Index (HI) developed by Hamzani & Chaushu (2018) and Landry (1988). The HI score ranges from 0 to 5, where 0 indicates poor healing and 5 indicates excellent healing.
  To ensure consistency and reliability in the assessment of healing, two independent researchers will evaluate the healing progress for all participants. The level of agreement between the researchers will be assessed using Cohen's Kappa index (Mandrekar, 2011). A Cohen's Kappa index value of 0.91 was achieved for the assessment of inflammation level, indicating a high degree of agreement. Similarly, agreement levels exceeding 0.90 were obtained across all HI levels, demonstrating a high level of concordance in the assessment of healing progress.
Post-surgical complications evaluated by presence or absense | 24 hours, 48 hours, 72 hours, and 7 days
  Monitoring and recording of any complications following the extraction procedure, such as alveolitis, trismus, infection, and hematoma (presence/absence).
  The presence of complications is related to a worse prognosis.
Oral Health-related Quality of Life measured by OHIP-14 test | 24 hours, 48 hours, 72 hours, and 7 days
  Assessment of the impact of treatment on patients' quality of life using validated instruments (OHIP-14).
  Lower scores: They indicate that the person experiences less impact of oral health problems on their quality of life. That is, they have fewer problems or feel less the impact of these problems in their daily lives.
  Intermediate scores: Suggest a moderate impact of oral health problems on quality of life. The person may experience some difficulties or discomfort related to their oral health, but they do not necessarily significantly affect their daily functioning.
  Higher scores: Indicate a significant impact of oral health problems on quality of life. The person may experience a wide range of problems that affect their general well-being, including pain, eating difficulties, sleep problems, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Abel García García, PhD, MD, Study Director — Universidade de Santaiago de Compostela
Locations (2):
- Spain (2):
  - Faculty of Dentistry of Universidade de Santiago de Compostela, Santiago de Compostela, A Coruña
  - Faculty of Dentistry University of Murcia, Murcia

IPD SHARING:
Plan to Share IPD: No